CLINICAL TRIAL: NCT06478849
Title: Adherence to and Understanding of a Therapeutic Education Program for Patients With Central Venous Lines
Brief Title: Adherence and Understanding of a Therapeutic Education Program for Patients With Central Venous Access (EDUVVC)
Acronym: EDUVVC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231313
Record Dates: First submitted 2024-06-03; First posted 2024-06-27 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-09

CONDITIONS: Therapeutic Education Program; Prevention
Keywords: central venous line
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: QUESTIONNAIRES — QUESTINNAIRES / WEBINARS
  Other Names: WEBINARS

SUMMARY:
The aim of this project is to evaluate, in a prospective cohort of PICC line patients, adherence to the project and understanding of the messages.

The transmission of knowledge and the acquisition of skills by patients with this type of invasive device will enable them to play an active role in their own care, and could help to reduce the frequency of risks.

This project is part of a collaborative approach that includes the creation of a mobile application for therapeutic education and monitoring (application under development). The evaluation of the device will be the subject of a national PHRC with national structures (SPIADI and PRIMO). The aim is to create a city-hospital collaboration to improve risk management.

DETAILED DESCRIPTION:
The ever-increasing use of central venous lines, including PICC lines, and the shift in medical practice towards ambulatory care, are making it increasingly complex to prevent the infectious and non-infectious risks associated with their use.

The involvement of numerous healthcare professionals within and outside the hospital, with varying levels of training, exposes patients to numerous complications, the incidence of which, depending on the device, ranges from 6 to 16%, and occur at the time of insertion (hematoma, pneumothorax, necrosis) or during use (infection, thrombosis, extravasation).

The transmission of knowledge and the acquisition of skills by patients wearing this type of invasive device helps to make the patient a player in his or her own care, and could help to reduce the frequency of risks. As part of a therapeutic education program, we aim to validate the communication tools and messages identified by a panel of French experts. These messages, together with the article published by Petit et al, have enabled us to draw up a skills reference framework for patients with a PICC line.

The aim of this project is to evaluate adherence to the project and understanding of the messages on a prospective cohort of patients.

This project is part of a collaborative approach that includes the creation of a mobile application for therapeutic education and monitoring (application under development). The evaluation of the device will be the subject of a national PHRC with national structures (SPIADI and PRIMO). The aim is to create a city-hospital collaboration to improve risk management.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 18 years of age
2. Patients requiring a PICC line
3. Patients with a means of communication with an Internet connection (computer or cell phone) or an alternative solution (landline telephone)
4. Patients with a predicted life expectancy of more than 6 weeks

Exclusion Criteria:

1. Patient opposed to participating in the study
2. Patient does not understand French
3. Patient not affiliated to a French social security scheme
4. Patient under guardianship or curatorship
5. Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with recent PICC line insertion, followed at AVICENNE hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-09-06 (Estimated); Study Completion 2025-10-21 (Estimated)

PRIMARY OUTCOMES:
Assess patients' level of understanding of communication tools. | WEEK 6 POST INCLUSION
  The level of comprehension will be assessed on the acquisition of the main messages and will be expressed as a percentage of correct answers.

SECONDARY OUTCOMES:
Estimating patient adherence to communication tools | WEEK 6 POST INCLUSION
  Adherence to communication tools will be assessed by the frequency of participation in the various webinars proposed.
Identify individual factors : a- Demographic b- Related to underlying pathology c- Management-related | week 6 post inclusion
  age, gender, ethnic origin, mother language, lifestyle, place of residence...

CONTACTS AND LOCATIONS:
Overall Officials: CAMILLE REINPRECHT, Principal Investigator — Hopital AVICENNE
Locations (1):
- Hopital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: No